CLINICAL TRIAL: NCT02597452
Title: Clinical Utility Study of a Low-Cost Hand-Held Breast Scanner
Acronym: iBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: UE LifeSciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 821412-UPCC24114
Record Dates: First submitted 2015-10-23; First posted 2015-11-05 (Estimated); Results first posted 2020-04-06 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer
Keywords: breast lump; breast exam; breast cancer screening; breast lump detection
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- intelligent Breast Exam, iBE (Other): Single Arm: Additional breast exam by a FDA approved hand-held intelligent breast exam device and a clinical breast exam during their scheduled breast screening appointment. No return visit required for participation.
  Interventions: Device: intelligent Breast Exam, iBE

INTERVENTIONS:
Device: intelligent Breast Exam, iBE — A bilateral iBE exam will be performed on the entire breast in addition to a clinical breast exam administered by a trained individual. If the patient is selected to participate in the inter-rater reliability portion of the study, the subject will undergo both the iBE and the clinical breast exams twice sequentially performed by two different separately trained individuals during the same visit.

SUMMARY:
The primary purpose of this study is to measure the clinical utility (accuracy) of the hand-held breast scanner (iBE) for the detection of breast lesions or lumps. The iBE results will be compared to the results of a current mammogram and/or ultrasound. The duration of study participation is approximately 30 minutes one day.

DETAILED DESCRIPTION:
The FDA approved class II device in this clinical trial is a low-cost hand-held breast scanner (intelligent Breast Exam, iBE). This device is to be used a pre-screening tool for mammograms or ultrasounds. Determination of the accuracy of iBE for the detection of clinically relevant breast lesions will be performed by means of a prospective study.

The iBE evaluation will be performed by a trained licensed practical nurse or ultrasound technologist who is blinded to the outcome of the radiology studies at the time the iBE is performed. The iBE training will be done by the leading iBE user in the United States. The iBE evaluation will be done prior to the patient's original scheduled imaging visit. After the completion of the imaging visit the radiologist will evaluate the mammogram and/or ultrasound images along with the iBE report.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Women and men with symptomatic breast lump (either by palpation or imaging) OR
* Asymptomatic women presenting to the imaging center for a screening mammogram
* Signed Informed Consent

Exclusion Criteria:

* Patients under 18 years of age
* Patients who previously participated in this study and are returning to the Women's Imaging Center for follow-up diagnostic tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2014-03; Primary Completion 2017-11-01 (Actual); Study Completion 2017-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ari D Brooks, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Pennsylvania Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Clanahan JM, Reddy S, Broach RB, Rositch AF, Anderson BO, Wileyto EP, Englander BS, Brooks AD. Clinical Utility of a Hand-Held Scanner for Breast Cancer Early Detection and Patient Triage. JCO Glob Oncol. 2020 Feb;6:27-34. doi: 10.1200/JGO.19.00205. PMID 32031433

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intelligent Breast Exam, iBE
Started | 516
Completed | 486
Not Completed | 30
Not completed — testing incomplete | 30

BASELINE CHARACTERISTICS:
Population: Patients analyzed were those who completed all exams required by the protocol.
Arm/Group | Intelligent Breast Exam, iBE
Number analyzed (Participants) | 486
Age, Continuous [Mean (Full Range); unit: years] | 58 [30 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 486
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 468
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 153
  White | 312
  More than one race | 2
  Unknown or Not Reported | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 486

OUTCOME MEASURES:

1. Primary Outcome: Compare the Outcomes of the iBE Examinations to Clinical Breast Examinations (CBE)by Estimating the Sensitivity of the Device Using Imaging Results
Description: comparing the calculated the sensitivities or the percentage of true positive breast lesions (based on imaging results) of the iBE and CBE
Time Frame: approximately one month after imaging scan
Measure: Number; unit: percentage of true positive lesions
Arm/Group | Intelligent Breast Exam, iBE
Number analyzed (Participants) | 486
percentage of true positive lesions | 34.3

2. Primary Outcome: Compare the Outcomes of the iBE Examinations to Clinical Breast Examinations by Estimating the Specificity of the Device Using Imaging Results
Description: comparing the calculated the specificities or the percentage of true negative lesions (based on imaging results) of the iBE and CBE
Time Frame: approximately one month after imaging
Measure: Number; unit: percentage of true negative lesions
Arm/Group | Intelligent Breast Exam, iBE
Number analyzed (Participants) | 486
percentage of true negative lesions | 80.3

3. Secondary Outcome: Position of the Breast Lesion as Measured by iBE and Mammography
Description: agreement of the position of the lesion, defined by time coordinate measured by iBE and mammography or ultrasound that fall within a 3 hour time quadrants on a clock of each other.
Time Frame: approximately one month after imaging
Population: Number of subjects who had a lesion identified by iBE and mammogram, ultrasound, or MRI.
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Intelligent Breast Exam, iBE
Number analyzed (Participants) | 5
Number analyzed (lesions) | 4
lesions | 4

4. Secondary Outcome: Size Detection of the Breast Lesions Identified by iBE
Description: The size detected of the breast lesion (cm) by mammogram or ultrasound
Time Frame: approximately one month after imaging
Population: The size was not measured by iBE. Only 4 of the 7 lesions were detected by iBE and size data was not available to analyze.
Units Other Than Participants: lesions
Arm/Group | Intelligent Breast Exam, iBE
Number analyzed (Participants) | 0
Number analyzed (lesions) | 0

5. Secondary Outcome: Inter-rate Reliability of the iBE and the CBE Number of Lesions Detected
Description: comparing the number of breast lesions detected two independent healthcare professionals consecutive evaluations of the same patient with the iBE device and clinical breast exam
Time Frame: through study completion an average of 18 months
Population: Difficulty enrolling patients for this outcome as a result of the participants undergoing the iBE and CBE twice by two different healthcare professionals. Subjects declined to continue after first healthcare professional exams was complete. Comparison data between healthcare professionals was not available to analyze.
Arm/Group | Intelligent Breast Exam, iBE
Number analyzed (Participants) | 0

6. Secondary Outcome: Inter-rate Reliability of the iBE and the CBE Position of Lesions Detected
Description: comparing the position(s) results of two independent healthcare professionals consecutive evaluations of the same patient with the iBE device and clinical breast exam
Time Frame: through study completion an average of 18 months
Population: as for outcome 5
Arm/Group | Intelligent Breast Exam, iBE
Number analyzed (Participants) | 0

7. Secondary Outcome: Post-stratification of the Analysis of the Reliability by Breast Imaging Reporting and Data System Level
Description: breakdown of the iBE clinically relevant findings and negative findings by the BIRAD levels determination from the gold standard final results
Time Frame: through study completion an average of 18 months
Population: The specificity of iBE relevant findings (BIRADs 0, 3-5) vs benign findings (BIRADS 1, 2) from the results of mammography
Measure: Count of Participants; unit: Participants
Arm/Group | Intelligent Breast Exam, iBE
Number analyzed (Participants) | 486
Participants
  iBE true positive findings | 12
  iBE true negative findings | 362
  iBE false positive findings | 89
  iBE flase negative findings | 23

ADVERSE EVENTS:
Time Frame: All participants were monitored for adverse events during a single visit, up to 1 hour.
Arm/Group | Intelligent Breast Exam, iBE
All-Cause Mortality (participants affected / at risk) | 0/486
Serious Adverse Events (participants affected / at risk) | 0/486
Other Adverse Events (participants affected / at risk) | 0/486

LIMITATIONS AND CAVEATS:
* difficulty recruiting patients with positive mammograms as this was unknown at time of enrollment
* difficulty recruiting patients for dual study for the inter-reliability study due to the increase in their scheduled visit time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-09): https://cdn.clinicaltrials.gov/large-docs/52/NCT02597452/Prot_SAP_000.pdf